CLINICAL TRIAL: NCT05459402
Title: Divided or Single Exposure (DOSE) Study: Randomized Controlled Trial for Pain in Persons Receiving Methadone Treatment
Brief Title: Divided or Single Exposure (DOSE) Study
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00318642; 1R01DA056045 (NIH); 1R01DA056045-01 (NIH)
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Chronic Pain; Methadone
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Methadone

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled for a 14-week Phase II between-group intervention period followed by a 6-month follow-up period with once monthly visits. All participants will be transitioned from liquid to tablet methadone within a 1 to 2-week period before being randomized to treatment as usual versus split daily methadone dosing for a 12-week period. Participants will complete monthly follow-up visits during months 4 - 9.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be done to prevent biasing participants or staff about the suspected group assignments. Blinded medication doses will be over-encapsulated by the research pharmacy, which will manage all randomization and blinding. Participants will be informed as part of their enrollment that no increases in methadone dosing will be permitted during the active intervention period; dose decreases will be permitted if determined necessary for safety purposes by medical providers and any changes will be implemented in a double-blinded manner by the study pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): Participants in treatment as usual group will receive 100% active methadone in AM + placebo in PM.
  Interventions: Drug: Methadone (100% dose)
- Split-dosing (Experimental): Participants in split dosing group will receive 50% active methadone + placebo twice daily.
  Interventions: Drug: Methadone (50% dose)

INTERVENTIONS:
Drug: Methadone (100% dose) — Methadone for the treatment of opioid use disorder
  Arms: Treatment as Usual (TAU)
Drug: Methadone (50% dose) — Methadone for the treatment of opioid use disorder
  Arms: Split-dosing

SUMMARY:
This study will evaluate whether once versus twice daily dosing of methadone will be an effective method for managing comorbid pain and opioid use disorder.

DETAILED DESCRIPTION:
This study follows a successfully completed project (NCT03254043) to now pursue the investigators overarching goal of optimizing methadone dosing as a method for managing comorbid chronic pain and opioid use disorder (OUD) among persons receiving methadone for the treatment of OUD. Up to 62% of persons maintained on methadone for OUD experience clinically significant pain, versus 31% in the general population. Pain in methadone-maintained persons (MMP) is associated with poor OUD treatment outcomes and severe distress. No effective treatment for comorbid pain and OUD currently exists; though preclinical and human data suggest divided methadone dosing may be a more optimal strategy for managing pain than once daily dosing, this has never been empirically examined. This study will evaluate an intervention for comorbid chronic pain among MMP using a Phase II double-blind, randomized, placebo-controlled comparison of treatment as usual (TAU) versus split daily methadone dosing for 12-weeks. Methadone will be remotely managed via an electronic pillbox. Outcomes will include weekly assessments of pain and OUD outcomes, ecological momentary assessment of pain before and after dosing, and point-prevalence measures of laboratory-induced pain to explore mechanism of effects. If effective, this approach could transform the care of MMP with pain because it would be feasible to implement within the operational structure of a methadone clinic and would impose low provider burden. Results could provide a high magnitude treatment for the substantial number of MMP who experience daily pain with no reliable form of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or older
* Currently receiving methadone for treatment of OUD for >90 days and have been consuming the same dose for >30 days
* Have previously received a take-home dose of methadone as part of routine care
* Willing to comply with study schedule
* Report pain (specific definition blinded)
* Have a cellular phone or be willing to carry phone provided by the study during one phase of the study

Exclusion Criteria:

* Pregnant
* Presence of acute medical problem that requires immediate and intense medical management
* Presence of a serious and unstable mental illness that interferes with provision of voluntary informed consent and/or adherence to study visits
* Plans to leave methadone treatment during the study period
* Maintained on a dose of methadone that would prevent effective splitting of doses
* Currently receiving split doses of methadone
* Currently receiving treatment for pain for which the split-dosing of methadone is judged by medical staff to be contraindicated or otherwise interfere with study conduct or integrity
* Does not meet criteria for mild-severe disability (definition blinded)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in worst pain rating- past 24 hour as assessed by the Brief Pain Inventory scale | Week 1 up to week 12
  Using the Brief Pain Inventory rating of "Worst Pain" in the past 24 hours, rated on a scale of 1-10, collected once weekly during weeks 1 through 12 of the intervention.

SECONDARY OUTCOMES:
Change in Pain Tolerance Latency | Weeks 1, 6, and 12
  Time in seconds (0-300) to removal of hand from cold pressor measure of laboratory-induced pain, collected point-prevalence during weeks 1, 6, and 12 of the intervention.
Change in Pain Interference- past 7 days as assessed by Pain-related Disability Scale Total Score | Week 1 up to 12
  Past 7 day Pain-related Disability Scale Total Score (range 0-70), collected once weekly during weeks 1 through 12 of the intervention.
Change in Opioid Withdrawal Severity- past 24 hours as assessed by the Subjective Opioid Withdrawal Scale | Week 1 up to 12
  Past 24 hour total score (range 0-64) for the Subjective Opioid Withdrawal Scale (SOWS), collected once weekly during weeks 1 through 12 of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Dunn, PhD, M.B.A., Principal Investigator — University of Maryland; Denis Antoine, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Addiction Treatment Services (ATS), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No